CLINICAL TRIAL: NCT02003404
Title: Preliminary Study of Peel Force and Discomfort of Removal of Adhesive Barriers in Normal and Peristomal Skin
Status: Completed | Type: Observational
Sponsor: Hollister Incorporated (Industry)
Collaborators: Loyola University (Other)
Responsible Party: Sponsor
Other Study IDs: 5642-O; LUHSC IRB #: 205654091813 (Other: Hollister Incorporated)
Record Dates: First submitted 2013-11-20; First posted 2013-12-06 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-10

CONDITIONS: Dermatologic Complications
Keywords: ostomy appliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Abdominal Skin: Apply SoftFlex (standard wear commercial skin barrier), FlexWear (standard wear commercial skin barrier), and FlexTend (extended wear commercial skin barrier), material to non-peristomal abdominal skin.
  Interventions: Device: Control Abdominal Skin
- Peristomal Abdominal Skin: Apply SoftFlex, FlexWear and FlexTend barrier material to peristomal abdominal skin.
  Interventions: Device: Peristomal Abdominal Skin

INTERVENTIONS:
Device: Control Abdominal Skin — Three barrier materials will be peeled from abdominal skin after a set period at a set rate.
  Other Names: SoftFlex; FlexWear; FlexTend
  Groups: Control Abdominal Skin
Device: Peristomal Abdominal Skin — Three barrier materials will be peeled from abdominal skin after a set period at a set rate.
  Other Names: SoftFlex; FlexWear; FlexTend
  Groups: Peristomal Abdominal Skin

SUMMARY:
This purpose of this study is to look at three commercially available ostomy barriers on peristomal (around the stoma) skin. Repeated barrier application and removal over years causes changes to the skin that the investigators wish to investigate. The primary objective is to measure peel force on normal skin and peel force on peristomal skin, with the intent of determining if differences occur. The study hypotheses is that no differences exist.

DETAILED DESCRIPTION:
This is a single center, non-invasive exploratory study utilizing a sample of convenience. This study compares three commercially available barrier materials on peristomal skin and normal abdominal skin.

ELIGIBILITY:
Inclusion Criteria:

* Colostomy, Ileostomy, or Urostomy patients at least 6 months post-surgery
* Males or females, age 18 to 80 years old at the time of enrollment
* Body Mass Index (BMI) between 18 and 50
* Willing to have two approximately 5" x 5" areas of the abdomen trimmed with a surgical clipper -- one in a ring around the stoma, and one on the opposite side
* Willing to remain within the testing room for the duration of the study
* Willing to allow a third person in the room as a witness for the duration of the study
* Able to position oneself onto and off of the examining table without the assistance of the Investigator
* Willing to refrain from vigorous exercise for the duration of the study
* Willing to not take any anti-inflammatory medications (except for Tylenol/acetaminophen) starting 48 hours prior to the study and for the duration of the study
* Willing to bring an extra barrier and replace their barrier worn during the study.
* Willing to follow the protocol as demonstrated by signing the Informed Consent Form
* In the opinion of the Investigator or qualified site personnel is qualified to participate

Exclusion Criteria:

* Clinically significant diseases, which may or may not be confined to the testing site, that may contraindicate participation; including but not limited to psoriasis, eczema, atopic dermatitis, and active cancer
* Use of topical drugs on the application site within 1 month.
* Use of lotions, creams, powders or oils on the application site in the 24 hours prior to application
* Pregnancy, lactation or planning a pregnancy as determined by interview only
* Other medical conditions, for example uncontrolled diabetes, which in the Investigator's judgment, makes the subject ineligible or places the subject at undue risk
* Participation in any clinical test either using the abdomen as a test site or using systemic therapy within the previous thirty days
* Damaged skin or other skin conditions in or near test sites which includes sunburn, scars, numerous moles or other disfiguration of the test site
* Significant adipose tissue at the test site that would preclude adequate adhesion of the study devices
* Known allergy to any of the test materials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ostomates with a normal peristomal skin and normal ipsilateral abdominal skin
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Swan, MD, Principal Investigator — Loyola University
Locations (1):
- La Grange Center for Health, La Grange Park, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 17 participants wore all three barrier types on control area AND peristomal area NOT 34 participants in study only 17 participants in study.
Groups:
- Abdominal Skin Barrier Peel Force: Barrier materials were attached and peeled off control and peristomal abdominal skin.
  Three commercial barrier materials (SoftFlex, FlexWear and FlexTend) were peeled from control or peristomal abdominal skin after a set period at a set rate.
Period: Overall Study
Arm/Group | Abdominal Skin Barrier Peel Force
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Must have ostomy of any type.
Groups:
- Abdominal Skin Barrier Peel Force: Three commerical barrier materials, SoftFlex, FlexWear and FlexTend barrier were peeled from control or peristomal abdominal skin after a set period at a set rate.
Arm/Group | Abdominal Skin Barrier Peel Force
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Skin Barrier Peel Force
Description: Peel force of barrier materials, comparing peristomal skin to abdominal skin. A portable peel force analyser, previously validated, was used in the clinic to measure peel at 90 degrees to the plane of the body. Peel force was measured on peristomal skin and ipsilateral abdominal skin in the same subject.
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: grams
Groups:
- Control Abdominal Skin Barrier Peel Force: Three commerical barrier materials, SoftFlex, FlexWear and FlexTend FlexWear barrier were peeled from abdominal skin after a set period at a set rate.
- Peristomal Skin Barrier Peel Force: Three commerical barrier materials, SoftFlex, FlexWear and FlexTend FlexWear barrier were peeled from peristomal skin after a set period at a set rate.
Arm/Group | Control Abdominal Skin Barrier Peel Force | Peristomal Skin Barrier Peel Force
Number analyzed (Participants) | 17 | 17
grams | 150 (10) | 215 (15)

ADVERSE EVENTS:
Time Frame: 5 months. Period from Sept 1, 2013 to Jan 31, 2014.
Arm/Group | Control Abdominal Skin Barrier Peel Force | Peristomal Skin Barrier Peel Force
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
Small sample size may not be generalizable to the population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No